CLINICAL TRIAL: NCT00203034
Title: A Multicenter, US and Canada, Double Blind, Randomized, Placebo-Controlled, Parallel Group Study, for the Efficacy, Tolerability and Safety of Rasagiline Mesylate in Levodopa Treated Parkinson's Disease Patients With Motor Fluctuations
Brief Title: Multicenter Study of Rasagiline in Parkinson's Disease Patients Using Levodopa and Experiencing Motor Fluctuations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Siyu Liu, MD, PhD, VP I R&D, Head of Global Clinical Operations, Teva Branded Pharmaceutical Products IR&D
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TV-1012/133
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental 1 (Experimental): 0.5 mg rasagiline mesylate oral once daily
  Interventions: Drug: rasagiline mesylate
- Experimental 2 (Experimental): 1.0 mg rasagiline mesylate oral once daily
  Interventions: Drug: 1.0 mg rasagiline mesylate
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: rasagiline mesylate — 0.5 mg rasagiline mesylate oral once daily
  Arms: Experimental 1
Drug: 1.0 mg rasagiline mesylate — 1.0 mg rasagiline mesylate oral once daily
  Arms: Experimental 2
Other: Placebo — oral placebo once daily
  Arms: Placebo

SUMMARY:
Study for patients currently using Levodopa/Carbidopa who will be assigned to receive either Rasagiline or Placebo

ELIGIBILITY:
Inclusion Criteria:

Men and women with idiopathic Parkinson's disease whose diagnosis is confirmed by at least two of the cardinal signs (resting tremor, bradykinesia, rigidity) being present, without any other known or suspected cause of parkinsonism.

Subjects must experience levodopa related motor fluctuations averaging at least 2.5 hours daily in the OFF state.

Subjects must be taking optimized levodopa/carbidopa or levodopa /benserazide carbidopa/levodopa therapy (based on investigator's judgment), stable for at least 14 days prior to baseline. Subjects must be receiving at least 3 daily doses of levodopa, not including a bedtime dose.

Selegiline must be discontinued for at least 90 days prior to baseline.

Subject must be age 30 or older.

Subjects must be willing and able to give informed consent.

Exclusion Criteria:

Subjects with a clinically significant or unstable medical or surgical condition which would preclude safe and complete study participation. Such conditions may include cardiovascular, pulmonary, hepatic, renal, or metabolic diseases or malignancies as determined by medical history, physical exam, laboratory tests, chest x-ray, or ECG for Parkinson's disease [e.g., pallidotomy, thalamotomy, and deep brain stimulation (DBS)] within the 12 months preceding the Baseline visit.

Subjects who have undergone neurosurgical transplantation are excluded regardless of when the procedure(s) was performed. No programming changes are permitted in subjects who have undergone DBS.

Participation in a previous clinical trial of rasagiline. Concomitant therapy with MAO inhibitors, reserpine, methyldopa within the past three months, or treatment with an anti-emetic or neuroleptic medication with central dopamine antagonist activity with the past six months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2000-05; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean total daily "OFF" time | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ira Shoulson, MD, Principal Investigator — The Parkinson Study Group
Locations (4):
- United States (4):
  - Rush - Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Columbia - Presbyterian Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Baylor College of Medicine, Houston, Texas